CLINICAL TRIAL: NCT02861313
Title: Oral Health Related Quality of Life and Peri-implant Condition in Single Implant Mandibular Overdenture Retained by CM LOC Versus Ball Attachment: A Randomized Controlled Trial
Brief Title: Oral Health Related Quality of Life and Peri-implant Condition in Single Implant Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Abdelaal Mohammed, Assisstant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-07-175
Record Dates: First submitted 2016-07-29; First posted 2016-08-10 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Quality of Life; Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM LOC attachment (Experimental): CM LOC attachment other names: resin matrix attachment
  Interventions: Device: CM LOC attachment
- ball attachment (Active Comparator): ball attachment other names metallic ball attachment
  Interventions: Device: ball attachment

INTERVENTIONS:
Device: CM LOC attachment — CM LOC attachment
  Other Names: resin matrix attachment
  Arms: CM LOC attachment
Device: ball attachment — Ball attachment
  Other Names: metallic ball attachment
  Arms: ball attachment

SUMMARY:
Comparing the quality of life and periimplant condition around a single implant retained mandibular overdenture in two groups one will have a ball attachment and the other is having a (CM-LOC) one.

DETAILED DESCRIPTION:
Single implant retained mandibular overdenture is considered an economic and simple treatment modality for edentulous subjects. Resin matrix (CM LOC) is one of the low profile attachments which represent a promising retention values with subsequent improvement in chewing ability and in turns enhance patient quality of life.Oral health impact profile for edentulous patient (OHIP-EDENT) is more specific to edentulous subjects.

Peri-implant soft tissue health (bleeding, inflammation, etc...) is a valuable marker to implant success. The study will record different attachment influenced-tissue response and its relation to implant success and oral health related quality of life (OHRQOL)

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for implantation.
* Each patient has to perform both a random blood sugar and Glycosylated Hemoglobin analysis. Patients with a Glycosylated hemoglobin test HbA1c up to 8% and a normal blood sugar level (79 to 110) or controlled diabetic patients (90-130 fasting according to American Association of Diabetes) will be included.
* Sufficient bone width (≥ 6 mm) in the anterior region to place an implant. It could be either normally present or achieved by bone plateauing. This will be confirmed by cone beam computed tomographic (CBCT) scans.
* Residual bone height ranging from 11-20 mm with the lowest vertical height in the midline of the mandible not less than 13 mm This will be confirmed by the CBCT.
* Patients seeking to install a single symphyseal implant and for whom new dentures will be constructed.
* Patients, who are dissatisfied with the retention and stability of their technically satisfactory dentures.
* Patients, who already have existing maxillary and mandibular complete dentures, and after examination of the mandibular dentures, it is found that there are technical problems with regard to denture design and/or occlusion; then new maxillary and mandibular dentures will be fabricated
* All patients should have adapted to their dentures for at least six weeks before being included in the trial.
* Patients providing written informed consents to participate in the trial and this will be done before the scheduled date for implant installation.

Exclusion Criteria:

* Patients with a systemic or local contra-indication for implant placement.
* Satisfied patients with the retention of their mandibular denture as well as unsatisfied patients with their maxillary denture.
* Patient with a mandibular denture height less than 6 mm between the base of the denture and the incisal edge of the central incisors (as measured by a caliper) or with 12 mm crown height space as measured by a ruler from the incisal edge till the crest of the ridge. This will be done from a putty index of the diagnostic set up.
* Incompliant and not cooperative patients.
* Patients smoking more than 10 cigarettes per day.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
change in oral health related quality of life using (oral health impact profile edentulous) questionnaire (OHIP-EDENT) | from baseline up to 5 years
  likert scale from 0-4

SECONDARY OUTCOMES:
change in modified gingival index | from baseline up to 5 years
  score measurement from 0-4 where 0 is no inflammation and 4 is sever inflammation
change in plaque index | from baseline up to 5 years
  score measurement from 0-3 where 0 denotes absence of plaque, 3 abundant plaque
modified bleeding index | from baseline up to 5 years
  score measurement from 0-3 where 0 denotes no bleeding, 3 profuse bleeding

CONTACTS AND LOCATIONS:
Overall Officials: marwa AA mohammed, A lecturer, Principal Investigator — non affliated
Locations (1):
- Removable Prosthodontic Department, Faculty of Oral and Dental Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided